CLINICAL TRIAL: NCT02558530
Title: Rapid Resolution of Human Fatty Liver Disease, the Key to Obesity-related Morbidity and Mortality
Brief Title: Resolution of Liver Fat in Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Marja-Riitta Taskinen, Professor, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atkins
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low carbohydrate diet (Other): Isocaloric diet, <20 g carbohydrates per day
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet — Isocaloric, carbohydrate restricted diet 14 days

SUMMARY:
The major adverse health consequences of obesity occur only when non-alcoholic fatty liver disease (NAFLD) also develops. NAFLD is characterized by abnormal hepatic accumulation of triglycerides and other lipids. The first-line approach to NAFLD management is caloric restriction and weight loss, but these remain difficult to achieve. Little attention has been given to dietary carbohydrate restriction, despite recent reports showing that hepatic de novo lipogenesis, a process that converts dietary carbohydrates into fatty acids in the postprandial state, accounts for approximately 25% of liver triglyceride content in hyperinsulinemic subjects with NAFLD. For comparison, only 15% of the liver triglycerides were derived from dietary fatty acids in patients with NAFLD who had consumed a standardized 30% fat diet for four days before being assessed.

DETAILED DESCRIPTION:
To establish the time-course of hepatic fat loss in NAFLD subjects on a carbohydrate-restricted diet (<20 g/day), a serial assessments of liver fat during two week diet will be performed. Also, markers of lipid and insulin metabolism, liver function test and changes in gut microbiota during rapid metabolic improvement will be assessed.

The overall aim is to exploit this unique set of human material to determine the specific cellular and molecular pathways that are modified in the early stages of metabolic improvement and fatty liver regression.

ELIGIBILITY:
Inclusion Criteria:

* increased liver fat above 5 % in magnetic resonance spectroscopy
* body mass index 27-39.9 kg/m2

Exclusion Criteria:

* liver cirrhosis
* portal hypertension
* chronic liver disease other than NAFLD
* diabetes mellitus or other significant endocrine disease
* any medication acting on nuclear hormone receptors or inducing liver enzymes or self-administration of supplements other than calcium or vitamins/trace elements
* any significant cardiovascular co-morbidity
* history of non-compliance
* genotype (PNPLA3-MM and TM6SF2-TT) promoting liver fat accumulation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Liver fat percent by nuclear magnetic resonance imaging | 14 days
  Liver fat percent measured by nuclear magnetic resonance imaging

SECONDARY OUTCOMES:
De novo lipogenesis measured as Incorporation of new fatty acids (%) to very-low density lipoprotein triglycerides | 14 days
Gut microbiota measured as change in microbiome profile from baseline | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Riitta Taskinen, Professor, Principal Investigator — University of Helsinki
Locations (2):
- RPU Diabetes and Obesity, Biomedicum, Helsinki, Finland
- Wllenberg Laboratory, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mardinoglu A, Wu H, Bjornson E, Zhang C, Hakkarainen A, Rasanen SM, Lee S, Mancina RM, Bergentall M, Pietilainen KH, Soderlund S, Matikainen N, Stahlman M, Bergh PO, Adiels M, Piening BD, Graner M, Lundbom N, Williams KJ, Romeo S, Nielsen J, Snyder M, Uhlen M, Bergstrom G, Perkins R, Marschall HU, Backhed F, Taskinen MR, Boren J. An Integrated Understanding of the Rapid Metabolic Benefits of a Carbohydrate-Restricted Diet on Hepatic Steatosis in Humans. Cell Metab. 2018 Mar 6;27(3):559-571.e5. doi: 10.1016/j.cmet.2018.01.005. Epub 2018 Feb 15. PMID 29456073